CLINICAL TRIAL: NCT07182890
Title: Efficacy of Clostridium Butyricum in Alleviating Anxiety and Depression in Patients With Functional Dyspepsia：A Prospective, Double-Blind, Randomized, Placebo-Controlled Clinical Trial
Brief Title: Efficacy of Clostridium Butyricum in Alleviating Anxiety and Depression in Patients With Functional Dyspepsia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20252363-C-1
Record Dates: First submitted 2025-09-05; First posted 2025-09-19 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-09

CONDITIONS: Functional Dyspepsia; Probiotics; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — phosphatidyltransferase, Clostridium butyricum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The probiotic group (Experimental): Probiotic Group:
  Patients with postprandial distress syndrome (PDS) will receive Mosapride Citrate Tablets 5 mg three times daily, along with Clostridium butyricum 1260 mg twice daily.
  Patients with epigastric pain syndrome (EPS) will receive Esomeprazole Enteric-Coated Tablets 20 mg once daily, along with Clostridium butyricum 1260 mg twice daily.
  Interventions: Drug: Clostridium butyricum
- The placebo group (Placebo Comparator): Placebo Group:
  Patients with PDS will receive Mosapride Citrate Tablets 5 mg three times daily, plus a placebo identical in appearance and odor to Clostridium butyricum (with identical dosage and frequency).
  Patients with EPS will receive Esomeprazole Enteric-Coated Tablets 20 mg once daily, plus a placebo identical in appearance and odor to Clostridium butyricum (with identical dosage and frequency).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Clostridium butyricum — Patients with postprandial distress syndrome (PDS) will receive Mosapride Citrate Tablets 5 mg three times daily, along with Clostridium butyricum 1260 mg twice daily.
  Patients with epigastric pain syndrome (EPS) will receive Esomeprazole Enteric-Coated Tablets 20 mg once daily, along with Clostridium butyricum 1260 mg twice daily.
  Arms: The probiotic group
Drug: placebo — Patients with PDS will receive Mosapride Citrate Tablets 5 mg three times daily, plus a placebo identical in appearance and odor to Clostridium butyricum (with identical dosage and frequency).
  Patients with EPS will receive Esomeprazole Enteric-Coated Tablets 20 mg once daily, plus a placebo identical in appearance and odor to Clostridium butyricum (with identical dosage and frequency).
  Arms: The placebo group

SUMMARY:
Objective: This study aims to evaluate the effectiveness of Clostridium butyricum in improving anxiety and depression in patients diagnosed with functional dyspepsia according to the Rome IV criteria.

Methods: This trial plans to enroll 180 patients (90 per group). The study will employ a double-blind design. For patients diagnosed with FD according to the Rome IV criteria, in addition to conventional treatment (treated with Mosapride Citrate Tablets (Guangdong Anno Guocai) for Postmeal Discomfort Syndrome (PDS) and Esomeprazole Enteric Coated Tablets (Shijiazhuang Longze Pharmaceutical Guocai) for Upper Abdominal Pain Syndrome (EPS)), the experimental group was treated with Clostridium butyricum, while the control group received a placebo with the same appearance and odor.

The treatment intervention will last for 4 weeks. The main indicator of this experiment is the improvement of the Hospital Anxiety and Depression Scale (HADS score) after 4 weeks of treatment. The secondary indicators are the improvement rate of the overall treatment effectiveness evaluation questionnaire (OTE questionnaire), the improvement of the global overall symptom score (GOS score), the improvement of the simplified Nipin scale (SF-NDI), and the improvement of the Pittsburgh Sleep Index (PSQI) after 4 weeks of treatment. Upon completion of the trial, the patients' conditions will be re-evaluated, and treatment plans will be adjusted accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with functional dyspepsia (FD) according to the Rome IV criteria.
* Aged 18 to 80 years, regardless of gender.
* Hospital Anxiety and Depression Scale (HADS) score between 8 and 14.

Exclusion Criteria:

* Use of probiotics or antibiotics within one month prior to the trial.
* Use of psychoactive medications (including hypnotics, sedatives, anxiolytics, or antidepressants) within one month prior to the trial.
* Use of hormones, immunosuppressants, or cytotoxic agents within one month prior to the trial.
* Participation in any other clinical trial within one month prior to the study.
* Positive test for Helicobacter pylori (Hp) infection.
* Long-term use of traditional Chinese herbal medicine.
* Pregnancy or lactation.
* History of drug abuse.
* Comorbidities such as irritable bowel syndrome (IBS), gastroesophageal reflux disease (GERD), functional constipation (FC), or other significant conditions that may interfere with the trial-including severe hepatic, renal, respiratory, or autoimmune disorders; bleeding diatheses; psychiatric diseases; endocrine disorders; etc.
* History of major surgery or diagnosis of diabetes mellitus.
* Refusal to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 4 weeks
  Hospital Anxiety and Depression Scale (HADS) is divided into an anxiety subscale (7 questions) and a depression subscale (7 questions), with each subscale scoring 0-21 points. The higher the score, the more severe the patient's anxiety and depression.

SECONDARY OUTCOMES:
Overall Treatment Evaluation (OTE) questionnaire | 4 weeks
  The OTE questionnaire uses the question "How have your stomach symptoms been in the past week compared to the baseline period?" scored on a 7-point Likert scale, with options of "extremely improved," "improved," "slightly improved," "unchanged," "slightly aggravated," "aggravated," or "extremely aggravated." If the patient answers "extremely improved" or "improved," it is considered a response, otherwise it is considered an unresponsive.
Global Overall Symptom scale (GOS score) | 4 weeks
  The GOS score evaluates 10 types of gastrointestinal symptoms, with each symptom scoring 1-7 points and a total score of 10-70 points. The higher the score, the more severe the symptoms.
Short-form Nepean Dyspepsia Index (SF-NDI) | 4 weeks
  Use Short-form Nepean Dyspepsia Index (SF-NDI) to evaluate the quality of life of patients, which includes 10 questions. Each question scores 1-5 points. The higher the score, the worse the quality of life.
Pittsburgh Sleep Quality Index (PSQI) | 4 weeks
  Pittsburgh Sleep Quality Index (PSQI) is a self-assessment scale used to evaluate sleep quality within the past month. It contains 7 components, each scored on a scale of 0-3, with a final total score range of 0-21. The higher the score, the worse the sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Air Force Medical University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No